CLINICAL TRIAL: NCT04383756
Title: Utilization of Donor Whole Blood for Blood Transfusion in Deceased Donor Liver Transplantation
Status: Withdrawn | Phase: Early Phase 1 | Type: Interventional
Why Stopped: Study was never started
Sponsor: Vanderbilt University Medical Center (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: UDWBBT
Record Dates: First submitted 2020-05-07; First posted 2020-05-12 (Actual); Last update posted 2022-03-09 (Actual); Status verified 2020-05

CONDITIONS: Transfusion Related Complication; Liver Transplant

STUDY DESIGN:
Intervention Model Description: 20 recipients receive donor whole blood 20 historic match controls are compared to the 20 study participants
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Donor Blood (Experimental): Between 2-4 units of donor leukoreduced whole blood (each unit will contain up to 350mL) transfused as needed in Liver transplantation participants
  Interventions: Biological: Donor Blood
- Banked Blood (Active Comparator): Standard of Care - Up to 350mL Allogenic banked component blood transfusion in a 1:1:1 manner (packed red blood cells : plasma : platelets) transfused as needed in Liver transplantation participants
  Interventions: Biological: Banked Blood

INTERVENTIONS:
Biological: Donor Blood — Up to 4 units (each unit contains 350mL) of leukoreduced donor whole blood
  Arms: Donor Blood
Biological: Banked Blood — Up to 350mL of Allogenic banked component blood transfusion in a 1:1:1 manner (packed red blood cells : plasma : platelets)
  Arms: Banked Blood

SUMMARY:
We will study 40 matched patients. 20 patients will receive leukoreduced whole blood from the solid organ donor. These 20 patients will be compared to 20 historical matched controls with regards to allogenic blood product usage and other physiologic markers

ELIGIBILITY:
Inclusion Criteria:

* - Recipients 18 years or older.
* Deceased donor whole graft liver transplant recipients undergoing liver transplant starting 07/01/2020 and onwards at VUMC.
* ABO-matched recipient and donor.
* Donor Hb level >/= 8 g/dL
* Recipients with negative ABO antibody screen

Exclusion Criteria:

* - Pediatric recipient.
* HBS Antigen+ donors
* HCV NAT+ donors
* Donors of A2 blood type
* Donors on oral anticoagulants (except for aspirin) over the past 3 days before organ procurement

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2020-12 (Estimated); Primary Completion 2021-07 (Estimated); Study Completion 2021-07 (Estimated)

PRIMARY OUTCOMES:
Use of allogenic banked blood products | perioperative up to 72 hours post operative
  Measured by the number of allogenic banked blood products used
Economic cost | perioperative up to 72 hours post operative
  Total cost of perioperative transfusions

SECONDARY OUTCOMES:
Number of Serious Adverse Events (SAEs) | Baseline to discharge (approximately 4-5 days)
  Number of deaths, life-threatening events, hospitalizations, disabilities or permanent damage, or congenital anomalies

CONTACTS AND LOCATIONS:
Overall Officials: Clayne Benson, MD, Principal Investigator — Vanderbilt University Medical Center
Locations (1):
- Vanderbilt University Medical Center, Nashville, Tennessee, United States

IPD SHARING:
Plan to Share IPD: No